CLINICAL TRIAL: NCT00011921
Title: Phase III Randomized Trial of Sequential High-Dose Chemotherapy Versus Standard Chemotherapy for the Treatment of Small Cell Lung Cancer
Brief Title: Chemotherapy Followed by Peripheral Stem Cell or Bone Marrow Transplant Compared With Chemotherapy Alone in Treating Patients With Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: EBMT Solid Tumors Working Party (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068379; EBMT-RANDOM-ICE; EU-98001; NCI-V01-1645
Record Dates: First submitted 2001-03-03; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2003-03

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer; extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Carboplatin; Epirubicin; Etoposide; etoposide phosphate; Ifosfamide; Paclitaxel; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: epirubicin hydrochloride
Drug: etoposide
Drug: etoposide phosphate
Drug: ifosfamide
Drug: paclitaxel
Procedure: autologous bone marrow transplantation
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy with peripheral stem cell transplant or bone marrow transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known whether high-dose chemotherapy plus peripheral stem cell or bone marrow transplant is more effective than chemotherapy alone in treating small cell lung cancer.

PURPOSE: This randomized phase III trial is studying how well chemotherapy followed by peripheral stem cell or bone marrow transplant works compared to chemotherapy alone in treating patients with limited-stage or extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the overall survival of patients with limited or extensive stage small cell lung cancer treated with sequential high-dose ifosfamide, carboplatin, and etoposide phosphate followed by autologous peripheral blood stem cell or bone marrow transplantation versus standard ifosfamide, carboplatin, and etoposide.
* Compare the progression-free survival, time to treatment failure, and response rate in patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to disease stage (limited disease vs extensive disease with vs without liver metastases), performance status (0 vs 1), gender, LDH level (normal vs abnormal), and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive induction therapy comprising epirubicin IV over 4 hours on day 1 and paclitaxel IV over 3 hours on day 2. Treatment repeats every 21 days for a total of 2 courses. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 3 and continuing for 10 days or during course 2 until peripheral blood stem cell (PBSC) collection is completed. After completion of induction chemotherapy, autologous PBSCs or bone marrow is collected.

Within 28 days of the start of the second course of induction chemotherapy, patients receive high-dose ifosfamide IV over 17 hours, carboplatin IV over 3 hours, and etoposide phosphate IV over 3 hours on days 1-4. At 48 hours after completion of high-dose chemotherapy, patients undergo autologous PBSC or bone marrow transplantation and then receive G-CSF SC for 14 days. Treatment repeats every 28 days for 3 courses.

* Arm II: Patients receive ifosfamide IV continuously over 24 hours, carboplatin IV over 1 hour on day 1, and etoposide IV over 45 minutes on days 1 and 2. Treatment repeats every 28 days for 6 courses.

After completion of high-dose or standard chemotherapy, patients with limited disease or extensive disease in complete remission receive thoracic radiotherapy daily on days 1-5 for 6 weeks. All patients in complete remission receive prophylactic cranial radiotherapy daily on days 1-5 for 3 weeks.

Quality of life is assessed at baseline, at the beginning of courses 1 and 3 (high-dose chemotherapy) or courses 3 and 5 (standard chemotherapy), and then at 7, 12, and 18 months.

Patients are followed monthly.

PROJECTED ACCRUAL: A total of 430 patients (215 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed small cell lung cancer

  * Limited disease or extensive disease with no more than 2 metastatic sites
* No CNS metastasis

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,500/mm^3 OR
* Platelet count greater than 100,000/mm^3 OR
* Hemoglobin at least 10.0 g/dL

Hepatic:

* AST/ALT less than 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2.5 times ULN
* Bilirubin less than 2.5 times ULN

Renal:

* Creatinine clearance at least 60 mL/min
* No renal function that would preclude chemotherapy

Cardiovascular:

* No congestive heart failure
* LVEF at least 50%
* No cardiac function that would preclude chemotherapy

Other:

* No other malignancy within the past 3 years except for basal cell skin cancer or carcinoma in situ of the cervix
* No psychiatric disorder or any other disorder that would preclude study participation
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 1997-09

PRIMARY OUTCOMES:
Overall survival (OS) at 3 years

SECONDARY OUTCOMES:
Progression-free survival (PFS) at 3 years
Toxicity at 3 years
Quality of life (QOL) at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Serge Leyvraz, MD, Study Chair — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland